CLINICAL TRIAL: NCT05894343
Title: Long-term Follow-up of Glutamic Acid Decarboxylase Gene Transfer to the Subthalamic Nuclei in Participants With Parkinson's Disease
Brief Title: Long-term Follow-up of Glutamic Acid Decarboxylase (GAD) Gene Transfer in Parkinson's Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MeiraGTx, LLC (Industry)
Responsible Party: Sponsor
Organization: MeiraGTx UK II Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGT-GAD-026
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to the follow-up or active treatment group based on the group to which they were randomized in Study MGT-GAD-025.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Follow-up group (No Intervention): Participants who were randomized to immediate treatment in Study MGT-GAD-025 will transition directly to a long-term follow-up schedule to complete an additional 54 months of follow-up. All study participants are to be followed for 60 months after vector administration.
- Active treatment group (Experimental): Participants who were randomized to sham surgery in Study MGT-GAD-025 will transition to an active treatment schedule, including open-label bilateral treatment, upon confirmation of continued eligibility. Upon completion of the treatment period, participants will enter the long-term follow-up schedule to complete a total of 60 months of follow-up.
  Interventions: Genetic: AAV-GAD

INTERVENTIONS:
Genetic: AAV-GAD — Bilateral infusion of AAV-GAD
  Arms: Active treatment group

SUMMARY:
The objective of this study is to evaluate the long-term safety of AAV-GAD delivered bilaterally to the subthalamic nuclei (STN) in participants with Parkinson's disease.

DETAILED DESCRIPTION:
The duration of individual participation in this study will be approximately 54 months for participants who received AAV-GAD in Study MGT-GAD-025 and approximately 60 months for participants who received sham surgery in Study MGT-GAD-025.

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled in Study MGT-GAD-025.

Exclusion Criteria:

* None

Ages: 25 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with study drug-related adverse events and serious adverse events | From study start until Month 60 post treatment

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Yale University, New Haven, Connecticut
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Weill Cornell Medicine, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - West Virginia University, Morgantown, West Virginia